CLINICAL TRIAL: NCT06770062
Title: Multimodality Evaluation of Left Ventricular Remodeling In Mitral Regurgitation: A Pilot Study
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alex K. Bratt, Division Chair of Thoracic Radiology, Mayo Clinic
Other Study IDs: 24-009436
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Left Ventricular Systolic Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic severe primary mitral regurgitation: Adults with chronic severe primary mitral regurgitation undergoing robotic mitral annuloplasty at Mayo Clinic Rochester
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Each subject will receive two cardiac MRI scans (with and without contrast), one preoperative and another 6-12 months after. The duration of each MRI is approximately 45-60 minutes

SUMMARY:
The purpose of this research is to determine the feasibility of a larger, future study proposing a multimodal approach using cardiac CT and MRI to assess the risk of developing left ventricular (LV) systolic dysfunction in patients with mitral regurgitation (MR).

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Male or Female
* A diagnosis of severe chronic primary mitral regurgitation
* Undergoing isolated robotic mitral annuloplasty at Mayo Clinic Rochester
* Patients must have the ability to consent or have an appropriate representative available to do so.

Exclusion Criteria:

* Prior valve intervention,
* Concomitant valve surgery at the time of mitral annuloplasty (e.g. tricuspid annuloplasty, aortic valve replacement).
* Concomitant >= moderate regurgitation or stenosis in any other valve by preoperative echocardiography
* History of prior myocardial infarction
* History of cardiomyopathy unrelated to mitral regurgitation (e.g. dilated, hypertrophic, infiltrative)
* Pregnancy. Women of childbearing potential will be verbally screened by clinical staff during as part of routine pre-MRI evaluation. If a subject is unsure whether they could be pregnant, a negative pregnancy test will be performed prior to scanning.
* Implantable devices that would be a contraindication to MRI
* Severe allergy to gadolinium MRI contrast

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with chronic severe primary mitral regurgitation undergoing robotic mitral annuloplasty at Mayo Clinic Rochester
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 2 years
  Number of subjects consented to participate in study
Dropout Rate | 2 years
  Number of subjects to withdraw from study
Systolic Dysfunction | 2 years
  Number of subjects to experience postoperative systolic dysfunction, defined as Left ventricular ejection fraction (LVEF) < 50%

CONTACTS AND LOCATIONS:
Overall Officials: Arman Arghami, MD, MPH, Principal Investigator — Mayo Clinic; Alex Bratt, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States